CLINICAL TRIAL: NCT02628158
Title: Correlation of Postoperative Vision and Fundus Autofluorescence After Vitrectomy for Epiretinal Membrane
Brief Title: Fundus Autofluorescence After Vitrectomy for Epiretinal Membrane
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Professor of Ophthalmology, Kyorin University
Other Study IDs: Kyorineye019
Record Dates: First submitted 2015-12-06; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Epiretinal Membrane
Keywords: Epiretinal membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Vitrectomy with internal limiting membrane removal — Vitrectomy with removal of epiretinal membrane and internal limiting membrane

SUMMARY:
Fundus autofluorescence (FAF) at the macula originates from hyperfluorescence from retinal pigment epithelium (RPE) and blockage of hyperfluorescence by macular pigment. Investigators evaluate whether presence of FAF may correlate to the postoperative visual outcome for epiretinal membrane.

DETAILED DESCRIPTION:
92 eyes with epiretinal membrane were performed vitreous surgery, epiretinal membrane removal and internal limiting membrane (ILM) peeling. Presence of hyperfluorescence in FAF at the macular area and best-corrected visual acuity (BCVA) was evaluated preoperatively and at postoperative 1, 3, and 6 months with ultra-wide angle imaging.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients who underwent vitrectomy and internal limiting membrane removal for epiretinal membrane and had followed for more than 6 months.

Exclusion Criteria:

* The patients with follow-up less than 6 months.

Ages: 20 Years to 90 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with epiretinal membrane who underwent vitrectomy with epiretinal membrane and internal limiting membrane removal
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Visual acuity before and after surgery | Changes from baseline to 1, 3, 6 months
  Vision

SECONDARY OUTCOMES:
Presence of fluids autofluorescence at the macular area | Changes from baseline up to 6 months
  Fundus autofluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided